CLINICAL TRIAL: NCT07398456
Title: Smartphone-enabled Hybrid Identification of Early CoLorectal Disease Using Blood-Based Cancer Testing Across TeXas
Acronym: SHIELD-TX
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: IRB TBD
Record Dates: First submitted 2026-02-04; First posted 2026-02-10 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Colorectal Cancer (CRC) Screening
Keywords: blood-based screening test; cancer risk; colorectal cancer risk; circulating tumor DNA; cell-free DNA; colorectal cancer screening
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients testing positive via BBST will be randomized based on clinic location such that half of the patients receive the intervention and the other half do not.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- App Intervention (Experimental): Patients on the app intervention arm will receive educational messages via their healthcare portal smartphone app.
  Interventions: Other: Educational Information via Smartphone App
- Standard Support (No Intervention): Patients on the standard support arm who receive a positive blood test result and either do not access their healthcare portal smartphone app and/or do not schedule a colonoscopy within 2 weeks of the blood test result will receive the standard patient navigation support offered which typically includes explanation and education regarding their positive test result and referral to a gastroenterologist or other proceduralist for a colonoscopy.

INTERVENTIONS:
Other: Educational Information via Smartphone App — The educational messages will include information about the meaning of a positive test result, the patient's chances of having a CRC detected on colonoscopy, and the importance of early CRC detection.
  Arms: App Intervention

SUMMARY:
The goal of this prospective implementation study is to understand the impact of a blood-based screening test (BBST) for colorectal cancer (CRC) on patient acceptability of and adherence to CRC screening as well as the rate of follow-up BBST in those with negative BBST at a 1-year interval.

Additional aims include assessing the impact of digital patient navigation intervention on the rate of follow-up colonoscopy in individuals with positive BBST. Patients will be randomized into the non-intervention arm or the intervention with an app arm.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 45-84 years of age
* Considered by health-care providers to be "average risk" for CRC as determined by USPSTF guidelines
* If a patient opts for BBST, they are able and willing to provide blood samples per protocol
* Ability to understand and the willingness to participate in the study
* Must have been seen in HTPN clinic within the past 24 months from study activation
* Must have active MyBSW app portal account and/or establish account during study recruitment

Exclusion Criteria:

* Patients with a personal history of CRC
* Patients with a known high-risk family history of CRC precluding the patient from being average risk
* Patients with known diagnosis of inflammatory bowel disease or history of polyps
* Patients who are currently symptomatic for CRC such as: blood in the stool
* Patients with any known medical condition which, in the opinion of the investigator, should preclude enrollment into the study
* Have a recorded up to date CRC screening in the EMR (within 1 year for FIT, 3 years for mt-sDNA, 10 years for colonoscopy)
* Patients with a previous abnormal colonoscopy finding who are due for surveillance.

Ages: 45 Years to 84 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5500 (Estimated)
Dates: Start 2026-06 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Blood-Based Screening Test (BBST) Follow-Up | 1 year after initial result
  Assess the number of patients with a negative BBST result who accept and complete a follow-up BBST.

SECONDARY OUTCOMES:
Patient Screening Test Preference | 1 year
  Assess patient preference rates and test completion rates for stool tests, colonoscopy, and blood-based CRC screening modalities.
Screening Rates | 1 year
  Compare the overall screening rates in the study population to a historical cohort in which blood-based testing was not offered as an option.
Intervention Efficacy | 1 year
  Assess whether use of a digital patient navigation tool +/- traditional patient navigation leads to an increased rate of completion of colonoscopy in those with a positive blood or stool test.

OTHER OUTCOMES:
Baseline BBST Results | 1 year
  Number of positive and negative BBST results at baseline testing.
Follow-Up BBST Results | 1 year after initial result
  Number of positive and negative BBST results at follow-up test
BBST+ Follow-Up | 1 year
  Number of BBST positives who received follow-up colonoscopy
BBST+/Colonoscopy- Follow-Up | 1 year after negative colonoscopy
  Percentage of BBST-positive/colonoscopy-negative patients who accept and complete the follow-up BBST after negative colonoscopy.

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor University Medical Center, Baylor Charles A Sammons Cancer Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided